CLINICAL TRIAL: NCT05605015
Title: Wearable Technology for Personalised Physical Activity Feedback in Cardiac Patients: a Feasibility
Brief Title: Wearable Technology for Personalised Physical Activity Feedback in Cardiac Patients: a Feasibility Study
Acronym: ACTIVE-CR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Royal United Hospitals Bath NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Daniella Springett, Principal Investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTIVE-CR-V1
Record Dates: First submitted 2022-10-19; First posted 2022-11-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTIVE-CR INTERVENTION (Experimental): Participants will complete a 6-week remote, technology-based physical activity intervention named ACTIVE-CR, in which they will be required to wear a wrist worn monitor to measure daily physical activity. Participants will be able to view their physical activity feedback on a web-based platform and will receive three online trainer sessions across the 6 weeks to help them to understand and interpret their data.
  Interventions: Behavioral: ACTIVE-CR
- CONTROL (No Intervention): Participants in the control group will receive usual care from their healthcare team (if relevant) and will be invited to have an assessment at baseline and 6-weeks. Control participants will not receive any form of intervention. At the end of the study, control participants will receive a summary of their physical activity data measured at baseline and 6-weeks (in a booklet format with guidance on how to interpret and use the information).

INTERVENTIONS:
Behavioral: ACTIVE-CR — The ACTIVE-CR intervention comprises three key components: a wrist-worn physical activity monitor, a web-based platform providing physical activity feedback, and three autonomy supportive online trainer sessions. Each component is grounded by multiple established behaviour change techniques consistent with the behaviour change taxonomy developed by Michie et al. (2013). The barriers to physical activity were identified in our previous work and are consistent with previous literature
  Arms: ACTIVE-CR INTERVENTION

SUMMARY:
Cardiac rehabilitation (CR) is a comprehensive, long-term secondary care programme offered to individuals after a heart attack to aid recovery and prevent further illness. If properly implemented, CR is highly effective at reducing cardiac mortality, re-event, and re-admissions. Despite the well-established benefits, less than 50% of eligible UK patients enrol on a CR program. Among those who do begin CR in the UK, drop-out rates of 12-55% have been reported. If the take up of CR were increased to 65% it would reduce readmissions by a third and save approximately £100 million per year.

Physical activity (PA) is the cornerstone of CR. With recent advances in wearable activity monitors, accurate and objective assessment of free-living PA is now possible. It is increasingly apparent that the health benefits of PA can be achieved in many ways, and multiple dimensions (or aspects) of PA are independently important. The most sophisticated wearable devices can be used to capture these different dimensions and provide a more comprehensive evaluation of free-living PA - enabling patients to understand their individual PA in the context of guidelines - and offering more behavioural options and personalised advice.

In prior work, the investigators have developed a digital system for patients to self-manage their PA. This system comprises a wearable wrist-mounted accelerometer, bespoke digital platform, plus remote virtual support. The digital system has been customised for CR based on qualitative research in cardiac patients and practitioners - who found PA feedback to be understandable and motivating - and a route to address barrier to taking part in CR. This study aims to examine the feasibility of delivering a 6-week trial of a remote, technology-enabled physical activity intervention to patients who were unable to take up or dropped out of CR in the last 12 months.

DETAILED DESCRIPTION:
Current provision of cardiac rehabilitation in the UK is only taken up by <50% of eligible patients, despite the importance of attending for managing symptoms, reducing hospital readmissions and mortality, and improving quality of life. Widely reported factors related to non-attendance include employment commitments, difficulties with transport, lack of time, distance to travel and embarrassment related to attending rehabilitation. The use of home-based programmes permits greater flexibility of CR delivery, as patients are able to complete their programme at a place and time that suit them, as well as increasing access for those who are unable to travel or do not live in close proximity to face-to-face classes. However, current home-based approaches are lacking in objective monitoring of patients and strategies to increase physical activity are limited, despite it being a core component of CR. It is increasingly apparent that the health benefits of physical activity can be achieved in many ways, and multiple dimensions (or aspects) of physical activity are independently important.

Our past research shows that many people misjudge their physical activity status because they do not have access to accurate personalised information. With recent advances in wearable activity monitors, accurate and objective assessment of daily physical activity is possible. The most sophisticated wearable devices can now be used to capture multiple dimensions of physical activity and thus improve the depth and quality of feedback provided to individuals. To date, technology-based physical activity interventions in CR have primarily targeted unidimensional physical activity outcomes, such as step counts and sedentary behaviour.

Multidimensional feedback provides greater awareness, insight, and a more complete understanding of personal physical activity; enabling individuals to take greater responsibility for managing their behaviour and in the context of physical activity guidelines. In addition, a multidimensional approach offers more behavioural options and personalised advice.

Therefore, this study aims to examine the feasibility of delivering a 6-week trial of a remote, technology-enabled physical activity intervention to patients who were unable to take up or dropped out of CR. This study addresses several further shortcomings of previous research in this area: 1) the lack of grounding in psychological behaviour change theory, 2) the lack of objective monitoring for physical activity in CR, and 3) the need for support from practitioners and/or trainers to facilitate physical activity behaviour change.

ELIGIBILITY:
Inclusion Criteria: Patients will be recruited in line with British Association for Cardiovascular Prevention and Rehabilitation (BACPR) guidelines, which states that the following priority patient groups shall be offered CR irrespective of age, sex, ethnic group, and clinical condition:

* Acute coronary syndrome
* Coronary revascularisation
* Heart failure

Other patient groups known to benefit:

* Stable angina
* Peripheral arterial disease
* Post-cerebrovascular event
* Post-implantation of cardiac defibrillators and resynchronisation devices
* Post-heart valve repair/replacement
* Post-heart transplantation and ventricular assist devices
* Adult congenital heart disease

Participants must also:

* Have access to a smart phone or tablet and the internet
* Have declined or dropped out of CR in the last 12 months

Exclusion Criteria: Patients who were not referred/deemed eligible for CR (assessed by clinical care team)

* No access to the internet and/or a smart phone
* Individuals who have completed CR in the last 12 months
* Unable to read English
* Unable to understand written or verbal information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: study recruitment | 6-weeks
  Assess recruitment rates, defined as the proportion of eligible patients who accept the invitation to participate in the study.
Feasibility: retention | 6-weeks
  Examine retention and adherence: defined as the proportion of participants who complete the study
Feasibility: adherence | 6-weeks
  Examine adherence: defined as the proportion of online trainer sessions completed and platform usage
Feasibility: acceptability | 6-weeks
  Explore the acceptability of the ACTIVE-CR intervention (in terms of affective attitude, burden, perceived effectiveness, ethicality, intervention coherence, opportunity costs, and self-efficacy) using The Theoretical Framework of Acceptability (TFA) Questionnaire

SECONDARY OUTCOMES:
Seven day physical activity measurement using a research grade device | 6-weeks
  A wrist worn physical activity monitor will be used to quantify the following physical activity measures derived from energy expenditure: sedentary time, and light, moderate, vigorous and very vigorous intensities of activity
Weight | 6-weeks
  Kilograms
Height | 6-weeks
  Centimetres
Waist circumference | 6-weeks
  Centimetres
Systolic and diastolic blood pressure | 6-weeks
  Measured in millimetres of mercury (mmHg)
Cholesterol levels (Low-density lipoproteins, high-density lipoproteins, total cholesterol) | 6-weeks
  Measured in millimoles per litre of blood
Triglyceride levels | 6-weeks
  Measured in millimoles per litre of blood
Functional capacity | 6-weeks
  Measured by the 6-minute walk test (metres)
Hospital Anxiety and Depression Scale | 6-weeks
  Score 0-7 represents "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe."
Dartmouth COOP Functional Assessment Charts | 6-weeks
  Overall quality of life, physical function, social function, pain. 9 questions, each with answers ranging from 1-5. Possible scores 9-45. The higher the score, the worse the outcome
Behavioural Regulation in Exercise Questionnaire-3 | 6-weeks
The Exercise Self-Efficacy Scale | 6-weeks
  Rating of participant's degree of confidence to 18 statements by recording a number from 0 to 100% for each one. The higher the score, the higher the degree of confidence.
International Physical Activity Questionnaire | 6-weeks
  Self-report measure for physical activity
Health Care Climate Questionnaire (short-form) | 6-weeks
  6 items, used to assess participant's perceptions of the degree to which their trainer was autonomy supportive. The scale ranges from 1-7 (scores therefore range from 6-42). The higher the score, the better the participant's perception of support from the trainer

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Peacock, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No